CLINICAL TRIAL: NCT00629356
Title: Follow-up the Health Condition , Investigation of the Immuno-regulation , and the Study for Interaction of Viral Hepatitis--- Among Patients With or After Dengue Fever Infection
Status: Withdrawn | Type: Observational
Why Stopped: The study had been revised and made a new application.
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Jih Jin Tsai/Dr, Kaoshing Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUH-IRB-960195
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2010-05

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: dengue fever

SUMMARY:
Originally test host's to understand the tracking healthily and immune change of the dengue fever in Taiwan. Blood drawing 20 c.c for liver examination, kidney and other biochemical function, analyze host immunity adjusts and controls the gene, and the reciprocation that may be produced with the virus hepatitis, besides collected 10 c.c urine at the same time. Urine check is in order to compare acute infect and infected over three month person, the change of chemical composition.

This plan expect to collect 150 healthy, 150 dengue fever infected and 150 dengue fever bleed hot or dengue fever shock disease group's patient, goal to understand health state and immunity of follow-up adjust and control the difference of the gene and the reciprocation may produce to virus hepatitis of light disease and serious disease.

DETAILED DESCRIPTION:
The dengue fever is an important tropical infectious disease in the south of Taiwan, cause and threaten of public health at Kaohsiung and Ping-Dong all over the years, this will cause patient's death, the default of clinical change of dengue fever, acute infect, infect influence, host immunity adjust and control, and the reciprocation of virus hepatitis, will be a very urgent in basic research.

Originally test host's to understand the tracking healthily and immune change of the dengue fever in Taiwan. Blood drawing 20 c.c for liver examination, kidney and other biochemical function, analyze host immunity adjusts and controls the gene, and the reciprocation that may be produced with the virus hepatitis, besides collected 10 c.c urine at the same time.

This plan expect to collect 150 healthy, 150 dengue fever infected and 150 dengue fever bleed hot or dengue fever shock disease group's patient, goal to understand health state and immunity of follow-up adjust and control the difference of the gene and the reciprocation may produce to virus hepatitis of light disease and serious disease.

Urine check is in order to compare acute infect and infected over three month person, the change of chemical composition. The result of study can help doctor to understand the factor of immune regulation and control of the host and health change after the dengue fever is infected with, possible reciprocation with virus hepatitis. Researchers have collect 100 dengue fever bleed hot or dengue fever shock syndrome groups of patient, it is estimated that can collect and expect the case will be counted within two years.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Dengue Fever

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patients who are suspicious of dengue infection.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-07; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Follow-up the Health Condition , Investigation of the Immuno-regulation , and the Study for Interaction of Viral Hepatitis--- Among Patients With or After Dengue Fever Infection

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Jin Tsai, MD, Study Director — Chung-Ho Memorial Hospital,Kaoshing Medical University
Locations (1):
- Kaoshing Medical University Chung-Ho Memorial Hospital, Kaoshiung, Taiwan